CLINICAL TRIAL: NCT03210558
Title: Effects of Moderately Increased Testosterone Concentration on Physical Performance and Behaviour in Healthy Women - a Double-blind, Randomized, Placebo-controlled Study
Brief Title: Study of Testosterone and Athlete Response
Acronym: STAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: The Swedish School of Sport and Health Sciences (Other)
Responsible Party: Principal Investigator, Angelica Lindén Hirschberg, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2016/1485-32
Record Dates: First submitted 2017-06-30; First posted 2017-07-07 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Athletic Performance; Testosterone; Women's Health: Female Athlete/Female Athlete Triad
Keywords: female athletes, testosterone, physical performance, body composition
MeSH Terms: conditions — Female Athlete Triad Syndrome

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized, placebo-controlled, phase II trial of in total 50 women randomized to two parallel groups (1:1): Group A treated with transdermal testosterone or Group B treated with placebo for ten weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The testosterone cream and the placebo cream will be of identical appearance and will have the same texture to maintain double blind treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Testosterone cream 1% (Andro-Feme® )
  Interventions: Drug: Testosterone cream 1% (Andro-Feme® )
- Group B (Placebo Comparator): Placebo cream
  Interventions: Drug: Placebo cream

INTERVENTIONS:
Drug: Testosterone cream 1% (Andro-Feme® ) — Testosterone cream 10 mg (1 ml) daily, supplied every evening via a dose applicator to the upper outer thigh for 10 weeks.
  Arms: Group A
Drug: Placebo cream — Placebo cream (1 ml) daily, supplied every evening via a dose applicator to the upper outer thigh for 10 weeks.
  Arms: Group B

SUMMARY:
Trial objectives and purpose: The primary aim is to study the effects of moderately increased testosterone concentration on aerobic performance (endurance running time to exhaustion), and secondary aims to investigate the effects on submaximal work on treadmill, anaerobic capacity, muscle strength, body composition, behaviour and well-being, blood parameters, steroid hormone profile, gynecological parameters and skeletal muscle parameters in young healthy women in a double-blind, randomized, placebo-controlled trial.

Treatment: Ten weeks of transdermal treatment with testosterone cream 10 mg daily or placebo cream in a randomized design (1:1).

Primary outcome: Aerobic performance (running time to exhaustion on treadmill)

Secondary outcomes:

1. Submaximal work on treadmill (oxygen uptake, ventilation, heart rate, blood lactate and subjective rate of exhaustion)
2. Anaerobic performance (Wingate test)
3. Muscle strength (Cybex apparatus, force transducer, counter movement jump)
4. Body composition (Dual X-ray Absorptiometry: muscle mass, fat mass, bone mass)
5. Behaviour and well-being (Quality of life, Profile of mood state, Confidence Questionnaire, Aggression Questionnaire)
6. Blood parameters (hemoglobin, hematocrit, reticulocytes, ferritin, CRP)
7. Steroid hormone profile in blood and urine
8. Gynecological evaluation (ovarian and endometrial variables on ultrasound)
9. Skeletal muscle morphology, metabolic enzymes and muscle protein synthesis

Study population: Fifty healthy menstruating women will be included in the study and randomized to treatment with testosterone or placebo. Inclusion criteria: 18-35 yrs of age; body mass index (BMI) 19-25; non-smoking; a moderate to high self-reported level of recreational physical activity; not taking hormonal contraception and willing to use highly efficient non-hormonal contraception during the study (intrauterine device, bilateral tubal occlusion, vasectomised partner, same-sex partner, or sexual abstinence); accepting to not participate in any sports competitive event during the study period plus one month. Exclusion criteria: the presence of cardiovascular, liver, biliary or renal disease; hyperlipidemia; uncontrolled high blood pressure; endocrinological disorder; oligomenorrhea (menstrual intervals of more than 6 weeks) or amenorrhea (no menstruation for at least 3 months); pregnancy; a history of thromboembolic disorder; any malignancy; and intake of hormonal contraception the last two months prior to the study.

ELIGIBILITY:
Inclusion criteria are: healthy menstruating women; 18-35 yrs of age; BMI 19-25; non-smoking; having a moderate to high self-reported level of recreational physical activity (minimum of three hours of endurance and/or strength training per week); not taking hormonal contraception; and willing to use highly efficient non-hormonal contraception during the study such as:

* Intrauterine device
* Bilateral tubal occlusion
* Vasectomised partner
* Same-sex partner
* Sexual abstinence

Exclusion criteria are: the presence of cardiovascular, liver, biliary or renal disease; hyperlipidemia; uncontrolled high blood pressure; endocrinological disorder; oligomenorrhea (menstrual intervals of more than 6 weeks) or amenorrhea (no menstruation for at least 3 months); pregnancy; a history of thromboembolic disorder; any malignancy; and intake of hormonal contraception the last two months prior to the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2018-06-20 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Aerobic performance | Baseline and 10 weeks of treatment
  Change in endurance exercise time to exhaustion on treadmill

SECONDARY OUTCOMES:
Submaximal work on treadmill | Baseline and 10 weeks of treatment
  Change in oxygen uptake (L/min, mL/kg x min)
Anaerobic performance (Wingate test) | Baseline and 10 weeks of treatment
  Change in average power output on a cycle ergometer (W)
Muscle strength (knee extension torque) | Baseline and 10 weeks of treatment
  Change in peak muscle strength (N) and strength endurance (time)
Functional power development-jump tests | Baseline and 10 weeks of treatment
  Change in jump height (m) by squat jump and countermovement jump
Physical activity during one week before treatment and one week before the end of treatment | Baseline and 10 weeks of treatment
  Change in accelerometer counts
Muscle mass | Baseline and 10 weeks of treatment
  Change in muscle mass (g) by DXA
Body fat percentage | Baseline and 10 weeks of treatment
  Change in body fat (%) by DXA
Bone mineral density | Baseline and 10 weeks of treatment
  Change in bone mineral density (g/cm2) by DXA
Psychological General Well-Being | Baseline and 10 weeks of treatment
  Change in Psychological General Well-Being (PGWB) score 0 (poor quality of life) and 110 (good quality of life)
Mood | Baseline and 10 weeks of treatment
  Change in mood (POMS) score 0 (not at all) to 4 (very much)
Confidence | Baseline and 10 weeks of treatment
  Change in confidence (Confidence Questionnaire) score 1 (not at all) to 5 (very much)
Aggression | Baseline and 10 weeks of treatment
  Change in aggression (Aggression Questionnaire) score 1 (does not fit in with me at all) to 5 (totally fits in with me)
Blood parameters | Baseline and 10 weeks of treatment
  Change in blood parameters (hemoglobin, hematocrit, reticulocytes, ferritin, CRP)
Steroid hormone profile in blood and urine | Baseline and 10 weeks of treatment
  Change in steroid hormones and metabolites in blood (testosterone, dihydrotestosterone, androstenedione, estradiol, dehydroepiandrosterone and its sulfate, cortisol, progesterone, other reproductive hormones (LH, FSH, AMH), binding protein (SHBG) and steroid hormones and metabolites in urine (estrone, estrone sulfate, androsterone glucuronide, 5α androstane-3α, 17β-diol 17-glucuronide, androst-5-ene-diol-3β, 17β-diol, testosterone, androstenedione, epitestosterone, androsterone, etiocholanolone).
Gynecological evaluation | Baseline and 10 weeks of treatment
  Change in ultrasound assessments of the endometrium (mm) and ovaries (volume)
Skeletal muscle | Baseline and 10 weeks of treatment
  Change in morphology and concentration of metabolic enzymes (HAD, SC), markers of muscle protein synthesis (mTOR, p70), as well as markers from the muscle atrophy pathway (MABbx, MuRF-1)

CONTACTS AND LOCATIONS:
Overall Officials: Angelica Lindén Hirschberg, Principal Investigator — Department of Obstetrics and Gynecology, Karolinska University Hospital, Stockholm, Sweden
Locations (1):
- Department of Obstetrics and Gynecology, Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bermon S, Ritzen M, Hirschberg AL, Murray TH. Are the new policies on hyperandrogenism in elite female athletes really out of bounds? Response to "out of bounds? A critique of the new policies on hyperandrogenism in elite female athletes". Am J Bioeth. 2013;13(5):63-5. doi: 10.1080/15265161.2013.776129. No abstract available. PMID 23557056
- [Background] Bermon S, Garnier PY, Hirschberg AL, Robinson N, Giraud S, Nicoli R, Baume N, Saugy M, Fenichel P, Bruce SJ, Henry H, Dolle G, Ritzen M. Serum androgen levels in elite female athletes. J Clin Endocrinol Metab. 2014 Nov;99(11):4328-35. doi: 10.1210/jc.2014-1391. Epub 2014 Aug 19. PMID 25137421
- [Background] Buss AH, Perry M. The aggression questionnaire. J Pers Soc Psychol. 1992 Sep;63(3):452-9. doi: 10.1037//0022-3514.63.3.452. PMID 1403624
- [Background] Chang WY, Knochenhauer ES, Bartolucci AA, Azziz R. Phenotypic spectrum of polycystic ovary syndrome: clinical and biochemical characterization of the three major clinical subgroups. Fertil Steril. 2005 Jun;83(6):1717-23. doi: 10.1016/j.fertnstert.2005.01.096. PMID 15950641
- [Background] Davis S, Papalia MA, Norman RJ, O'Neill S, Redelman M, Williamson M, Stuckey BG, Wlodarczyk J, Gard'ner K, Humberstone A. Safety and efficacy of a testosterone metered-dose transdermal spray for treating decreased sexual satisfaction in premenopausal women: a randomized trial. Ann Intern Med. 2008 Apr 15;148(8):569-77. doi: 10.7326/0003-4819-148-8-200804150-00001. PMID 18413618
- [Background] Davis SR, Hirschberg AL, Wagner LK, Lodhi I, von Schoultz B. The effect of transdermal testosterone on mammographic density in postmenopausal women not receiving systemic estrogen therapy. J Clin Endocrinol Metab. 2009 Dec;94(12):4907-13. doi: 10.1210/jc.2009-1523. Epub 2009 Oct 22. PMID 19850682
- [Background] El-Hage G, Eden JA, Manga RZ. A double-blind, randomized, placebo-controlled trial of the effect of testosterone cream on the sexual motivation of menopausal hysterectomized women with hypoactive sexual desire disorder. Climacteric. 2007 Aug;10(4):335-43. doi: 10.1080/13697130701364644. PMID 17653960
- [Background] Fenichel P, Paris F, Philibert P, Hieronimus S, Gaspari L, Kurzenne JY, Chevallier P, Bermon S, Chevalier N, Sultan C. Molecular diagnosis of 5alpha-reductase deficiency in 4 elite young female athletes through hormonal screening for hyperandrogenism. J Clin Endocrinol Metab. 2013 Jun;98(6):E1055-9. doi: 10.1210/jc.2012-3893. Epub 2013 Apr 30. PMID 23633205
- [Background] Fooladi E, Reuter SE, Bell RJ, Robinson PJ, Davis SR. Pharmacokinetics of a transdermal testosterone cream in healthy postmenopausal women. Menopause. 2015 Jan;22(1):44-9. doi: 10.1097/GME.0000000000000259. PMID 24845394
- [Background] Goldstat R, Briganti E, Tran J, Wolfe R, Davis SR. Transdermal testosterone therapy improves well-being, mood, and sexual function in premenopausal women. Menopause. 2003 Sep-Oct;10(5):390-8. doi: 10.1097/01.GME.0000060256.03945.20. PMID 14501599
- [Background] Gooren LJ, Bunck MC. Transsexuals and competitive sports. Eur J Endocrinol. 2004 Oct;151(4):425-9. doi: 10.1530/eje.0.1510425. PMID 15476439
- [Background] Hagmar M, Berglund B, Brismar K, Hirschberg AL. Hyperandrogenism may explain reproductive dysfunction in olympic athletes. Med Sci Sports Exerc. 2009 Jun;41(6):1241-8. doi: 10.1249/MSS.0b013e318195a21a. PMID 19461542
- [Background] Meriggiola MC, Jannini EA, Lenzi A, Maggi M, Manieri C. Endocrine treatment of transsexual persons: an Endocrine Society Clinical Practice Guideline: commentary from a European perspective. Eur J Endocrinol. 2010 May;162(5):831-3. doi: 10.1530/EJE-09-1091. Epub 2010 Feb 11. PMID 20150325
- [Background] Huang G, Basaria S, Travison TG, Ho MH, Davda M, Mazer NA, Miciek R, Knapp PE, Zhang A, Collins L, Ursino M, Appleman E, Dzekov C, Stroh H, Ouellette M, Rundell T, Baby M, Bhatia NN, Khorram O, Friedman T, Storer TW, Bhasin S. Testosterone dose-response relationships in hysterectomized women with or without oophorectomy: effects on sexual function, body composition, muscle performance and physical function in a randomized trial. Menopause. 2014 Jun;21(6):612-23. doi: 10.1097/GME.0000000000000093. PMID 24281237
- [Background] Jovanovic H, Kocoska-Maras L, Radestad AF, Halldin C, Borg J, Hirschberg AL, Nordstrom AL. Effects of estrogen and testosterone treatment on serotonin transporter binding in the brain of surgically postmenopausal women--a PET study. Neuroimage. 2015 Feb 1;106:47-54. doi: 10.1016/j.neuroimage.2014.11.003. Epub 2014 Nov 11. PMID 25462800
- [Background] Mooradian AD, Morley JE, Korenman SG. Biological actions of androgens. Endocr Rev. 1987 Feb;8(1):1-28. doi: 10.1210/edrv-8-1-1. PMID 3549275
- [Background] Notelovitz M. Androgen effects on bone and muscle. Fertil Steril. 2002 Apr;77 Suppl 4:S34-41. doi: 10.1016/s0015-0282(02)02968-0. PMID 12007900
- [Background] Rickenlund A, Carlstrom K, Ekblom B, Brismar TB, von Schoultz B, Hirschberg AL. Hyperandrogenicity is an alternative mechanism underlying oligomenorrhea or amenorrhea in female athletes and may improve physical performance. Fertil Steril. 2003 Apr;79(4):947-55. doi: 10.1016/s0015-0282(02)04850-1. PMID 12749436
- [Background] Slayden SM. Risks of menopausal androgen supplementation. Semin Reprod Endocrinol. 1998;16(2):145-52. doi: 10.1055/s-2007-1016265. PMID 9711680
- [Background] Turpeinen U, Linko S, Itkonen O, Hamalainen E. Determination of testosterone in serum by liquid chromatography-tandem mass spectrometry. Scand J Clin Lab Invest. 2008;68(1):50-7. doi: 10.1080/00365510701496496. Epub 2007 Jun 24. PMID 17852804
- [Background] Zang H, Carlstrom K, Arner P, Hirschberg AL. Effects of treatment with testosterone alone or in combination with estrogen on insulin sensitivity in postmenopausal women. Fertil Steril. 2006 Jul;86(1):136-44. doi: 10.1016/j.fertnstert.2005.12.039. Epub 2006 Jun 5. PMID 16750207
- [Background] Zang H, Sahlin L, Masironi B, Eriksson E, Linden Hirschberg A. Effects of testosterone treatment on endometrial proliferation in postmenopausal women. J Clin Endocrinol Metab. 2007 Jun;92(6):2169-75. doi: 10.1210/jc.2006-2171. Epub 2007 Mar 6. PMID 17341565
- [Background] Zethraeus N, Kocoska-Maras L, Ellingsen T, von Schoultz B, Hirschberg AL, Johannesson M. A randomized trial of the effect of estrogen and testosterone on economic behavior. Proc Natl Acad Sci U S A. 2009 Apr 21;106(16):6535-8. doi: 10.1073/pnas.0812757106. Epub 2009 Apr 6. PMID 19366676
- [Derived] Horwath O, Moberg M, Hirschberg AL, Ekblom B, Apro W. Molecular Regulators of Muscle Mass and Mitochondrial Remodeling Are Not Influenced by Testosterone Administration in Young Women. Front Endocrinol (Lausanne). 2022 Apr 14;13:874748. doi: 10.3389/fendo.2022.874748. eCollection 2022. PMID 35498440
- [Derived] Elings Knutsson J, Andersson A, Baekken LV, Pohanka A, Ekstrom L, Hirschberg AL. Disposition of Urinary and Serum Steroid Metabolites in Response to Testosterone Administration in Healthy Women. J Clin Endocrinol Metab. 2021 Mar 8;106(3):697-707. doi: 10.1210/clinem/dgaa904. PMID 33274381
- [Derived] Hirschberg AL, Elings Knutsson J, Helge T, Godhe M, Ekblom M, Bermon S, Ekblom B. Effects of moderately increased testosterone concentration on physical performance in young women: a double blind, randomised, placebo controlled study. Br J Sports Med. 2020 May;54(10):599-604. doi: 10.1136/bjsports-2018-100525. Epub 2019 Oct 15. PMID 31615775